CLINICAL TRIAL: NCT02615795
Title: Tele Health Monitoring Service for Patients With Chronic Obstructive Pulmonary Disease. A Clinical, Randomized, Controlled Study for Evaluation of Clinical and Economic Consequences of Monitoring Service
Brief Title: Tele Health Monitoring Service for Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UAarhusFA
Record Dates: First submitted 2015-11-18; First posted 2015-11-26 (Estimated); Last update posted 2019-10-02 (Actual); Status verified 2010-10

CONDITIONS: Chronic Obstructive Pulmonary Disease, COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Best practice
- Intervention (Experimental): Best practice + Tele Monitoring of physiological parameters (heart frequence, oxygen saturation, weight, FEV1), and answers to disease specific questions, using Tunstall monitoring device.
  Interventions: Device: Tele Monitoring, using Tunstall monitoring device

INTERVENTIONS:
Device: Tele Monitoring, using Tunstall monitoring device — Monitoring of symptoms and physiological parameters at home, using Tunstall Healthcare telemedicine equipment. Patients perform physiological measurement. In addition, they correspond to a standardized questionnaire regarding disease specific symptoms. Data is assessed by the medical staff the same day. If the data indicates worsening in the patient's condition, the patient is contacted by phone. The assessment of the patient is made either on the specialist nurse level, or at a conference between the specialist nurse and a senior pulmonary doctor. There is no call center service.
  Other Names: Tunstall monitoring device
  Arms: Intervention

SUMMARY:
The aim of this study is to evaluate the effect of monitoring patients with chronic obstructive pulmonary disease (COPD) after a hospitalization for COPD exacerbation or pneumonia. The patients are randomized to receive either standard treatment and follow up, or standard treatment and follow up, plus tele monitoring of key clinical parameters and symptoms for six months.

DETAILED DESCRIPTION:
Telemedicine is a relatively new approach for the management of chronic obstructive pulmonary disease (COPD) disease. Telemedicine, for monitoring disease exacerbation, is the focus area of our research. The patient monitoring offers the possibility of early initiation of treatment of patients who has evidence of COPD exacerbation or pulmonary infection. The self-monitoring of potential exacerbation is started after a hospitalization, and is done by the patient on a daily (not on weekends) basis initially. After one month the monitoring is made at least three times weekly during the rest of the intervention period of six months. With the help of the monitoring equipment, the patient answers a short series of health related questions, and makes simple measurements of oxygen saturation, heart rate, lung function and weight. Data is sent to the hospital, and here the staff can assess the data and respond to them the same day, with a phone call to the patient, if the patient's condition has changed. The selected telemonitoring-equipment, consists of a monitoring systems for the assessment of key clinical parameters and symptoms. All patients, in the intervention group as well as in the control group, are trained in the use of a standardized self-treatment plan. It is expected that the monitoring of symptoms and signs will support patient empowerment.

The investigation is planned to assess the clinical and economic effects of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Obstructive Pulmonary Disease COPD with FEV1/FVC (Forced Expiratory Volume in 1 second / Forced Vital Capacity) below 70% at all times during the study. FEV1 below 51% during inclusion and during the further study. Inclusion takes place during a hospitalization, with exacerbation in pulmonary symptoms.

Exclusion Criteria:

* Not able to give written or oral consent
* Terminal disease, such as cancer
* Unstable heart disease, such as coronary infarction within the last to month
* Disabling psychiatric disease
* Asthma
* Inability to use the equipment
* Severe language barriers
* Drug abuse
* Alcohol abuse

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2011-03; Primary Completion 2018-06-06 (Actual); Study Completion 2018-06-06 (Actual)

PRIMARY OUTCOMES:
Number of hospitalization days | During twelve months

SECONDARY OUTCOMES:
Duration of COPD related hospitalizations, in days | Twelve months
Number of hospitalizations caused by COPD exacerbation | During twelve months
Number of COPD related contacts to emergency rooms | Twelve months
Number of self-addressed COPD exacerbations | Twelve months
  Without primary contact to medical staff
Sensitivity of physiological measurements in detecting COPD exacerbation | During six months of intervention
  Relation between physiological measurements and COPD exacerbation
Number of unplanned contact to primary health sector | Twelve months
  Contacts to general practitioner or Doctor on call in the primary health sector
Health related quality of life | Twelve months
  Saint George´s respiratory questionnaire, Hospital Anxiety and Depression score, SF-36 questionnaire
Number of all cause contacts to primary health sector | Twelve months
  Contacts to general practitioner or Doctor on call in the primary health sector
Mortality | During twelve months

CONTACTS AND LOCATIONS:
Overall Officials: Frank D Andersen, MD, Principal Investigator — Diagnostic Center, Regional Hospital of Silkeborg
Locations (1):
- Region Hospital of Silkeborg, Silkeborg, Mid Region, Denmark